CLINICAL TRIAL: NCT02640976
Title: Assessing the Relation Between Hormone Receptors Gene Polymorphism and Ovarian Stimulation Response in In Vitro Fertilization (IVF) Program
Brief Title: Poor Ovarian Stimulation Response in In Vitro Fertilization (IVF) Program
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadine wagdi maurice, Demonstrator at faculty of pharmacy Cairo university biochemistry department, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BC (705)
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: in vitro fertilization; controlled ovarian hyperstimulation; poor ovarian response; estrogen receptor 2 gene polymorphism; follicle stimulating hormone receptor gene polymorphism; anti-mullerian hormone
MeSH Terms: conditions — Infertility | interventions — Menotropins; hMG-IBSA; cetrorelix; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Poor responders (Active Comparator): This group will include women who underwent IVF/ICSI cycle and produced 4 oocytes or less.
  intervention:
  1. fixed daily morning dose of Human menopausal gonadotrophin (HMG) Merional® intra-muscular injection ,starting on cycle day 2 and will be maintained for 9-11 days according to each individual ovarian response,at a dose of (300 IU).
  2. On cycle day 7, the GnRH antagonist Cetrorelix 0.25 mg Cetrotide® will be introduced as daily subcutaneous injections and continued till the day of ovulation triggering.
  3. Finally, when at least 3 follicles will reach 17 mm in diameter, ovulation will be triggered by a single intra-muscular injection of 10,000 IU of Human chorionic gonadotrophin (hCG) Choriomon®.
  Interventions: Drug: Human menopausal gonadotrophin (HMG); Drug: GnRH antagonist Cetrorelix; Drug: Human chorionic gonadotrophin (hCG)
- Good responders (Active Comparator): This group will include women who produced (5 or more oocytes) after COH.
  Intervention:
  1. fixed daily morning dose of Human menopausal gonadotrophin (HMG) Merional® intra-muscular injection ,starting on cycle day 2 and will be maintained for 9-11 days according to each individual ovarian response,at a dose of (225 IU) for participants with AMH levels > 1.5 ng/ml and/or FSH levels ≤ 8 mIU/ml
  2. On cycle day 7, the GnRH antagonist Cetrorelix 0.25 mg Cetrotide® will be introduced as daily subcutaneous injections and continued till the day of ovulation triggering.
  3. When at least 3 follicles will reach 17 mm in diameter, ovulation will be triggered by a single intra-muscular injection of 10,000 IU of Human chorionic gonadotrophin (hCG) Choriomon®.
  Interventions: Drug: Human menopausal gonadotrophin (HMG); Drug: GnRH antagonist Cetrorelix; Drug: Human chorionic gonadotrophin (hCG)

INTERVENTIONS:
Drug: Human menopausal gonadotrophin (HMG) — [Merional® 75 IU ampoules, IBSA institut]
  Other Names: Merional®
Drug: GnRH antagonist Cetrorelix — [Cetrotide® 0.25 mg syringes, Merck Serono]
  Other Names: Cetrotide®
Drug: Human chorionic gonadotrophin (hCG) — [Choriomon® 5000 IU ampoules, IBSA institut]
  Other Names: Choriomon®

SUMMARY:
The aim of this study is to assess the role of AMH in prediction of poor ovarian response as well as the relation between ESR2 (+1730G>A) (rs4986938), FSHR p.Thr307Ala (c.919A>G, rs6165) and FSHR p.Asn680Ser (c.2039A>G, rs6166) SNPs and the poor response in Egyptian women undergoing IVF procedure. Discovering the genetic variants associated with ovarian response is an important step towards individualized pharmacogenetic protocols of ovarian stimulation.

DETAILED DESCRIPTION:
In-vitro fertilization treatment safety is highly challenged by the erratic individual variability to controlled ovarian hyperstimulation (COH). One of the diverse predictive factors is the AMH, which is considered to be the most sensitive marker. Nowadays, practices of pharmacogenetics could predict the stimulation success and thus tailoring the treatment reaching advancement in patient care. Since the efficiency of the Follicle stimulating hormone (FSH) dose is greatly related to the success of COH, the FSHR gene is treated as the primary candidate in explaining the difference in COH results.Furthermore, the estrogen receptors are important genes for improvements in the diagnosis and treatment of infertility.

Materials and Methods: Starting June 2013, couples with unexplained infertility, seeking the first attempt IVF/ICSI treatment cycle will be recruited in "AL shark Al-Awsat fertility center".In this prospective study, 216 Couples fulfilling our inclusion criteria will enroll in this study after informed consent. Ovarian stimulation will be performed according to the GnRH antagonist protocol with a fixed daily morning dose of Human menopausal gonadotrophin (HMG) [Merional® 75 IU ampoules, IBSA institut] intra-muscular injection starting on cycle day 2. Based on the patient's body mass index and hormonal profile, the daily dose of HMG will be adjusted to (225 IU) for participants with AMH levels > 1.5 ng/ml and/or FSH levels ≤ 8 mIU/ml and to (300 IU) for participants with AMH levels < 1.5 ng/ml and/or FSH levels > 8 mIU/ml, doses will be increased by 75 IU in cases with BMI > 30 Kg/m2. On day 2 of the menstrual cycle, the dose of HMG will be commenced for all patients and will be maintained for 9-11 days according to each participant individual ovarian response assessed by trans-vaginal ultrasound folliculometry starting on cycle day 7 and continued every other day until the day of Human chorionic gonadotrophin (hCG) injection. On cycle day 7, the GnRH antagonist Cetrorelix 0.25 mg [Cetrotide® 0.25 mg syringes, Merck Serono] will be introduced as daily subcutaneous injections and continued till the day of ovulation triggering. Finally, when at least 3 follicles will reach 17 mm in diameter, ovulation will be triggered by a single intra-muscular injection of 10,000 IU of hCG [Choriomon® 5000 IU ampoules, IBSA institut]. 36 hours later, oocyte retrieval will be performed and will be guided by transvaginal ultrasound. According to our primary outcome, the number of oocytes collected, patients will be classified as poor responders (4 oocytes or less) and will be considered as good responders if they produced 5 or more oocytes. The good responders group will serve as the control group.

Genotyping:Peripheral blood will be collected from each patient in an EDTA-containing tube. Genomic DNA will be extracted from lymphocytes of peripheral blood by fully automated system of QIAcube using QIAamp DNA Blood Mini Kit (250) plus QIAamp DNA Blood Mini Accessory Set B, cat. no. 1043369. Detection of the polymorphisms ESR2 (+1730G>A) (rs4986938), FSHR p.Thr307Ala (c.919A>G, rs6165) and FSHR p.Asn680Ser (c.2039A>G, rs6166) SNPs will be performed using the TaqMan system by real-time polymerase chain reaction (PCR). Primers and probes will be provided by applied biosystem, Life Technologies. Assays will be performed with TaqMan Universal Master Mix.

Statistical analysis: Data will be statistically described in terms of mean and standard deviation, for quantitative data and frequencies (number of cases) and relative frequencies (percentages) for qualitative data. Hardy-Weinberg (H-W) Equilibrium for each polymorphism will be tested using the Chi-square test. Comparison of quantitative variables will be done using unpaired t test when comparing 2 categories and one way analysis of variance (ANOVA) with post hoc test when comparing more than 2 categories.

For comparing categorical data, Chi square test will be performed. Exact test will be used instead when the expected frequency is less than 5.

Genotype and allele frequencies will be compared between the disease and the control groups using chi-square tests. Odds ratio (OR) with 95% confidence intervals will be calculated. A probability value (P value) less than 0.05 will be considered statistically significant. All statistical calculations will be done using SPSS (Statistical Package for the Social Science; SPSS Inc., Chicago, IL, USA) version 22.

ELIGIBILITY:
Inclusion Criteria:

* Women at or under the age of 35 years.
* Normal thyroid stimulating hormone and prolactin levels.
* Normal ovulatory cycles (25-35 interval days), together with proven patent fallopian tubes at hysterosalpingography or laparoscopy done within six cycles preceding the ICSI cycle.
* Presence of both ovaries with normal findings as assessed by trans-vaginal ultrasound and laparoscopy.
* All male partners had a normal semen analysis according to WHO criteria (WHO, 2010), done within 6 months preceding the ICSI cycle

Exclusion Criteria

* Chronic medical disorders such as diabetes.
* Previous inadequate response to ovulation induction.
* Polycystic ovary syndrome.
* Women who performed ovarian surgery and cases of endometriosis diagnosed by laparoscopy or suspected by ultrasound or CA-125 assay.
* Abnormal pelvic pathology or congenital anomalies.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
number of oocytes collected | 3 weeks from of start of ICSI cycle
  when at least 3 follicles will reach 17 mm in diameter, ovulation will be triggered by a single intra-muscular injection of 10,000 IU of hCG [Choriomon® 5000 IU ampoules, IBSA institut]. 36 hours later, oocyte retrieval will be performed and will be guided by transvaginal ultrasound.

SECONDARY OUTCOMES:
Detection of the single nucleotide polymorphisms ESR2(+1730G>A) (rs4986938), FSHR p.Thr307Ala (c.919A>G, rs6165) and FSHR p.Asn680Ser (c.2039A>G, rs6166) SNPs will be performed using the TaqMan system by real-time polymerase chain reaction (PCR) | Within 1 week
  By using PCR, we will indicate the genotype in each individual and determine the probability of the poor ovarian response.

OTHER OUTCOMES:
Laboratory analysis of basal follicle stimulating hormone level for each individual will be measured by enzyme-linked immunosorbent assay (ELISA) | Done within 3 months preceeding the ICSI cycle
  Based on FSH level, the dose of HMG ( Merional) will be adjusted for each individual.
Laboratory analysis of anti-mullerian hormone level (AMH) will be measured by ELISA technique for each individual. | Done within 3 months preceeding the ICSI cycle.
  Based on AMH level, the dose of HMG (Merional) will be adjusted for each individual.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Motawi TMK, Rizk SM, Maurice NW, Maged AM, Raslan AN, Sawaf AH. The role of gene polymorphisms and AMH level in prediction of poor ovarian response in Egyptian women undergoing IVF procedure. J Assist Reprod Genet. 2017 Dec;34(12):1659-1666. doi: 10.1007/s10815-017-1013-4. Epub 2017 Aug 19. PMID 28825151